CLINICAL TRIAL: NCT05257317
Title: Efficacy of Cranial Manual Therapy in the Treatment of Chronic Insomnia Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Escoles Universitaries Gimbernat (Other)
Collaborators: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Maider Sánchez Padilla, Principal Investigator, Escoles Universitaries Gimbernat
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019/302
Record Dates: First submitted 2022-01-24; First posted 2022-02-25 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Sleep Initiation and Maintenance Disorders
Keywords: Sleep Iniciation and Maintenane Disorders; Autonomic Nervous System; Osteopathic Medicine; Muskuloeskeletal Manipulation; Dysominias
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): It will consist of osteopathic manual therapy techniques applied to the occipital and temporal bones.
  Interventions: Other: Osteopathic Medicine
- Placebo (Placebo Comparator): It consists of a light contact applied to the cranial vault (frontal and parietal bones) where circular movements will be induced.
  Interventions: Other: Placebo therapy

INTERVENTIONS:
Other: Osteopathic Medicine — Where compression and traction movements will be carried out on these structures.
  Technique called CV4, applied on the occipital, and Technique called asynchronous rolling of the temporal bones.
  Arms: Intervention
Other: Placebo therapy — Circular movements will be induced in a frontal and parietal bones
  Arms: Placebo

SUMMARY:
Insomnia is the most prevalent sleep disorder in society. The first treatment of choice is pharmacology, although it can have secondary effects such as tolerance and dependence, or alter the structure of sleep; therefore, new pathways towards other adjuvant treatments are being established. OBJECTIVES: The main objective is "To assess the effectiveness of manual cranial therapy on the quantity and quality of sleep in patients with chronic insomnia." MATERIAL AND METHODS: A randomized clinical trial is designed, with two groups, intervention and placebo, to assess the effectiveness of manual therapy applied to the skull, in the severity of insomnia, and quantity and quality of sleep in patients with sleep disorder. chronic insomnia. Health professionals will be selected from the Department of Occupational Health, with characteristics of chronic insomnia described by the ICSD-III, who do not modify their usual medication regimen (if they take it) and without other pathologies related to sleep that may be causing the insomnia. insomnia Demographic data (age, sex, profession), clinical (BMI, history of previous and family insomnia pathologies, and taking medication for sleep and related disorders), sleep quality questionnaires (PSQI, COS, ISI) will be collected. , stress-insomnia relationship (FISRST-S), and quality of life (SF12), in addition to filling out a sleep diary (through the mobile App) and recording activity through actigraphy, hypnogram (Sleep ProfilerTM); before and after the intervention, and at one and three month follow-up. Each group will receive the offered intervention: cranial manual therapy (intervention) or cranial massage (placebo). The data will be coded and analyzed with the IBM SPSS® version 20 program (or similar)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with chronic insomnia disorder according to the criteria defined by the ICSD-III (International Classification of Sleep Disorders-3rd edition):

  * Problems initiating or maintaining sleep, associated with daytime consequences; and not attributable to environmental circumstances.
  * Insomnia lasting more than 3 months, with episodes of at least 3 times a week.
* Regarding the pharmacology or medication indicated for sleep:

  * They do not want to take the medication recommended by the doctor who is treating them.
  * Do not change their usual drug regimen, if they were already taking medication to sleep.
  * They are not taxed to take medication.
* Having ruled out other pathologies related to sleep through:

  * Respiratory polygraphy to rule out sleep-related respiratory pathologies (SAHS).
  * screening to rule out motor sleep disorders.
  * screening to rule out circadian sleep disorders.
  * screening to rule out serious psychiatric disorders (depression, anxiety, general psychopathology): BDI-II (Beck Depression Inventory), BAI (Beck Anxiety Inventory), SCL-90.
* Obtain a score greater than 7 points (clinical-subclinical insomnia).

Exclusion Criteria:

* Obtain a score of less than 7 (clinically insignificant insomnia) in the ISI test (Insomnia Severity Index).
* The result of the respiratory polygraphy is positive, confirming a sleep-disordered breathing.
* The screening tests for the detection of motor sleep disorders, respiratory sleep disorders or circadian disorders are positive.
* The Screening detects serious psychiatric illnesses such as major depressive disorder or bipolar disorders is positive.
* Suffering or having suffered from any central neurological pathology, stroke, aneurysm...
* Having suffered skull fractures.
* Having undergone surgery in the last 6 months and that insomnia has started as a result of it.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity | 18 weeks
  With an "Insomnia Severity Index" (ISI). There are seven items. Each item is rated on a scale from 0 to 4 from less to more severe. The total score is the sum of each individual item and can range from 0 to 28 (28 = most severe insomnia).

SECONDARY OUTCOMES:
Sleep Quality | 18 weeks
  With a "Pittsburgh Sleep Quality Index (PSQI)" It consists of 19 items that analyze: quality, latency, duration, efficiency and sleep disturbances, use of sleeping medication and daytime dysfunction. The scores of the questions allows between 0 and 3 points for each of the seven subscales, where in all cases a score of "0" indicates ease, while a score of "3" indicates severe difficulty within its respective area. The sum of the seven subscales allows obtaining a global score between 0 and 21 for the entire scale, where "0" indicates ease of sleeping and "21" severe difficulty in all areas.
Sleep Quality | 18 weeks
  With a "Cuestionario del Sueño de Oviedo (COS)". It consists of 15 items, 13 of which are grouped into 3 scales:
  * Subjective sleep satisfaction (1 item): score from 1 to 7.
  * Insomnia (9 items) The scoring range is from 9 to 45, higher score indicate greater severity.
  * Hypersomnia (3 items): from 3 to 15 points, higher score indicate greater daytime disability.
Vulnerability to stress-related insomnia | 9 weeks
  With FORD INSOMNIA RESPONSE TO STRESS spanish (FIRST-S). It is a scale that assesses vulnerability to stress-related insomnia. It is a standardized questionnaire with high test-retest reliability, which has been validated as a predictive measure of sleep vulnerability using polysomnographically measured sleep. It is made up of nine items and requires the individual to rate between 1 (not at all common) and 4 (very common) the probability of having sleep disturbance in association with specific and common stressful events or periods of stress that occur during the day or at night .
  The total score of the answers obtained is quantified. High scores are indicative of increased vulnerability to stress-related insomnia. The cut-off score to detect individuals with this vulnerability is 19 points or higher, indicating "high-FIRST sleep reactivity."
Quality of Life of patients with insomnia | 18 weeks
  With a 12-items Short-Form Health Survey (SF12). It consists of 12 items from the 8 dimensions of the SF-36 Physical Function (2), Social Function (1), Physical Role (2), Emotional Role (2), Mental Health (2), Vitality (1), Body Pain (1), General Health (1). The response options form Likert-type scales that assess intensity or frequency. The number of response options ranges from three to six, depending on the item.
  For each of the 8 dimensions that it identifies, the items are coded, aggregated and transformed into a scale ranging from 0 (the worst state of health for that dimension) to 100 (the best state of health).
Quantity, latency and efficiency of sleep | 18 weeks
  With a "Sleep Diary"
Quantity, latency and efficiency of sleep | 18 weeks
  With an "Actigraphy record"
Hypnogram-Polysomnography - Macro and microstructure of sleep | 18 weeks
  With a "WachPAt(R) device"
Heart Rate Variability | 4 weeks
  With a "Polar H10 band" and "EliteHRV" app

CONTACTS AND LOCATIONS:
Overall Officials: Maider Sánchez-Padilla, MSc, Principal Investigator — Escoles Universitaries Gimbernat; Laura Vigil-Gimenez, PhD, Study Director — Corporación Parc Taulí; Maria José Masdeu-Margalef, PhD, Study Director — Corporación Parc Taulí
Locations (1):
- Escoles Universitaries Gimbernat, Sant Cugat del Vallès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
The pandemic has delayed the completion of the study and no publication date for the information has been proposed

REFERENCES:
- [Background] Equihua-Benitez AC, Guzman-Vasquez K, Drucker-Colin R. Understanding sleep-wake mechanisms and drug discovery. Expert Opin Drug Discov. 2017 Jul;12(7):643-657. doi: 10.1080/17460441.2017.1329818. Epub 2017 May 22. PMID 28511597
- [Background] Riemann D, Spiegelhalder K, Feige B, Voderholzer U, Berger M, Perlis M, Nissen C. The hyperarousal model of insomnia: a review of the concept and its evidence. Sleep Med Rev. 2010 Feb;14(1):19-31. doi: 10.1016/j.smrv.2009.04.002. Epub 2009 May 28. PMID 19481481
- [Background] Durmer JS, Dinges DF. Neurocognitive consequences of sleep deprivation. Semin Neurol. 2005 Mar;25(1):117-29. doi: 10.1055/s-2005-867080. PMID 15798944
- [Background] Riemann D, Nissen C, Palagini L, Otte A, Perlis ML, Spiegelhalder K. The neurobiology, investigation, and treatment of chronic insomnia. Lancet Neurol. 2015 May;14(5):547-58. doi: 10.1016/S1474-4422(15)00021-6. Epub 2015 Apr 12. PMID 25895933
- [Background] Merino-Andreu M, Alvarez-Ruiz de Larrinaga A, Madrid-Perez JA, Martinez-Martinez MA, Puertas-Cuesta FJ, Asencio-Guerra AJ, Romero Santo-Tomas O, Jurado-Luque MJ, Segarra-Isern FJ, Canet-Sanz T, Gimenez-Rodriguez P, Teran-Santos J, Alonso-Alvarez ML, Garcia-Borreguero Diaz-Varela D, Barriuso-Esteban B. [Healthy sleep: evidence and guidelines for action. Official document of the Spanish Sleep Society]. Rev Neurol. 2016 Oct 3;63(s02):1. Spanish. PMID 27699758
- [Background] Nofzinger EA, Buysse DJ, Germain A, Price JC, Miewald JM, Kupfer DJ. Functional neuroimaging evidence for hyperarousal in insomnia. Am J Psychiatry. 2004 Nov;161(11):2126-8. doi: 10.1176/appi.ajp.161.11.2126. PMID 15514418
- [Background] Halasz P, Bodizs R, Parrino L, Terzano M. Two features of sleep slow waves: homeostatic and reactive aspects--from long term to instant sleep homeostasis. Sleep Med. 2014 Oct;15(10):1184-95. doi: 10.1016/j.sleep.2014.06.006. Epub 2014 Jul 8. PMID 25192672
- [Background] Bastien CH, St-Jean G, Morin CM, Turcotte I, Carrier J. Chronic psychophysiological insomnia: hyperarousal and/or inhibition deficits? An ERPs investigation. Sleep. 2008 Jun;31(6):887-98. doi: 10.1093/sleep/31.6.887. PMID 18548835
- [Background] Sateia MJ. International classification of sleep disorders-third edition: highlights and modifications. Chest. 2014 Nov;146(5):1387-1394. doi: 10.1378/chest.14-0970. PMID 25367475
- [Background] Morgenthaler T, Alessi C, Friedman L, Owens J, Kapur V, Boehlecke B, Brown T, Chesson A Jr, Coleman J, Lee-Chiong T, Pancer J, Swick TJ; Standards of Practice Committee; American Academy of Sleep Medicine. Practice parameters for the use of actigraphy in the assessment of sleep and sleep disorders: an update for 2007. Sleep. 2007 Apr;30(4):519-29. doi: 10.1093/sleep/30.4.519. PMID 17520797
- [Background] Riha RL. Diagnostic approaches to respiratory sleep disorders. J Thorac Dis. 2015 Aug;7(8):1373-84. doi: 10.3978/j.issn.2072-1439.2015.08.28. PMID 26380763
- [Background] Thorpy MJ. Classification of sleep disorders. Neurotherapeutics. 2012 Oct;9(4):687-701. doi: 10.1007/s13311-012-0145-6. PMID 22976557
- [Background] D'Alonzo GE, Krachman SL. Circadian rhythm sleep disorders. J Am Osteopath Assoc. 2000 Aug;100(8 Suppl):S15-21. PMID 11002615
- [Background] Medrano-Martinez P, Ramos-Platon MJ. [Cognitive and emotional alterations in chronic insomnia]. Rev Neurol. 2016 Feb 16;62(4):170-8. Spanish. PMID 26860722
- [Background] Nijs J, Mairesse O, Neu D, Leysen L, Danneels L, Cagnie B, Meeus M, Moens M, Ickmans K, Goubert D. Sleep Disturbances in Chronic Pain: Neurobiology, Assessment, and Treatment in Physical Therapist Practice. Phys Ther. 2018 May 1;98(5):325-335. doi: 10.1093/ptj/pzy020. PMID 29425327
- [Background] Sateia MJ, Buysse DJ, Krystal AD, Neubauer DN, Heald JL. Clinical Practice Guideline for the Pharmacologic Treatment of Chronic Insomnia in Adults: An American Academy of Sleep Medicine Clinical Practice Guideline. J Clin Sleep Med. 2017 Feb 15;13(2):307-349. doi: 10.5664/jcsm.6470. PMID 27998379
- [Background] Riemann D, Voderholzer U, Spiegelhalder K, Hornyak M, Buysse DJ, Nissen C, Hennig J, Perlis ML, van Elst LT, Feige B. Chronic insomnia and MRI-measured hippocampal volumes: a pilot study. Sleep. 2007 Aug;30(8):955-8. doi: 10.1093/sleep/30.8.955. PMID 17702263
- [Background] Molen YF, Carvalho LB, Prado LB, Prado GF. Insomnia: psychological and neurobiological aspects and non-pharmacological treatments. Arq Neuropsiquiatr. 2014 Jan;72(1):63-71. doi: 10.1590/0004-282X20130184. PMID 24637973
- [Background] Kingston J, Raggio C, Spencer K, Stalaker K, Tuchin PJ. A review of the literature on chiropractic and insomnia. J Chiropr Med. 2010 Sep;9(3):121-6. doi: 10.1016/j.jcm.2010.03.003. PMID 22027034
- [Background] Benca RM. Diagnosis and treatment of chronic insomnia: a review. Psychiatr Serv. 2005 Mar;56(3):332-43. doi: 10.1176/appi.ps.56.3.332. PMID 15746509
- [Background] Schutte-Rodin S, Broch L, Buysse D, Dorsey C, Sateia M. Clinical guideline for the evaluation and management of chronic insomnia in adults. J Clin Sleep Med. 2008 Oct 15;4(5):487-504. PMID 18853708
- [Background] Ohayon MM. Epidemiology of insomnia: what we know and what we still need to learn. Sleep Med Rev. 2002 Apr;6(2):97-111. doi: 10.1053/smrv.2002.0186. PMID 12531146
- [Background] Morin CM, Benca R. Chronic insomnia. Lancet. 2012 Mar 24;379(9821):1129-41. doi: 10.1016/S0140-6736(11)60750-2. Epub 2012 Jan 20. PMID 22265700
- [Background] Ohayon MM, Sagales T. Prevalence of insomnia and sleep characteristics in the general population of Spain. Sleep Med. 2010 Dec;11(10):1010-8. doi: 10.1016/j.sleep.2010.02.018. Epub 2010 Nov 18. PMID 21093362
- [Background] Gronli J, Soule J, Bramham CR. Sleep and protein synthesis-dependent synaptic plasticity: impacts of sleep loss and stress. Front Behav Neurosci. 2014 Jan 21;7:224. doi: 10.3389/fnbeh.2013.00224. eCollection 2013. PMID 24478645
- [Background] Meerlo P, Koehl M, van der Borght K, Turek FW. Sleep restriction alters the hypothalamic-pituitary-adrenal response to stress. J Neuroendocrinol. 2002 May;14(5):397-402. doi: 10.1046/j.0007-1331.2002.00790.x. PMID 12000545
- [Background] Xie Z, Chen F, Li WA, Geng X, Li C, Meng X, Feng Y, Liu W, Yu F. A review of sleep disorders and melatonin. Neurol Res. 2017 Jun;39(6):559-565. doi: 10.1080/01616412.2017.1315864. Epub 2017 May 1. PMID 28460563
- [Background] Lomeli HA, Perez-Olmos I, Talero-Gutierrez C, Moreno CB, Gonzalez-Reyes R, Palacios L, de la Pena F, Munoz-Delgado J. Sleep evaluation scales and questionaries: a review. Actas Esp Psiquiatr. 2008 Jan-Feb;36(1):50-9. PMID 18286400
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] Dodds KL, Miller CB, Kyle SD, Marshall NS, Gordon CJ. Heart rate variability in insomnia patients: A critical review of the literature. Sleep Med Rev. 2017 Jun;33:88-100. doi: 10.1016/j.smrv.2016.06.004. Epub 2016 Jun 28. PMID 28187954
- [Background] Qaseem A, Kansagara D, Forciea MA, Cooke M, Denberg TD; Clinical Guidelines Committee of the American College of Physicians. Management of Chronic Insomnia Disorder in Adults: A Clinical Practice Guideline From the American College of Physicians. Ann Intern Med. 2016 Jul 19;165(2):125-33. doi: 10.7326/M15-2175. Epub 2016 May 3. PMID 27136449
- [Background] McCall WV. Cognitive behavioral therapy for insomnia (CBT-I): What is known, and advancing the science by avoiding the pitfalls of the placebo effect. Sleep Med Rev. 2018 Apr;38:1-2. doi: 10.1016/j.smrv.2017.05.001. Epub 2017 May 5. No abstract available. PMID 28655580
- [Background] Shergis JL, Ni X, Jackson ML, Zhang AL, Guo X, Li Y, Lu C, Xue CC. A systematic review of acupuncture for sleep quality in people with insomnia. Complement Ther Med. 2016 Jun;26:11-20. doi: 10.1016/j.ctim.2016.02.007. Epub 2016 Feb 18. PMID 27261976
- [Background] Bialosky JE, Bishop MD, Price DD, Robinson ME, George SZ. The mechanisms of manual therapy in the treatment of musculoskeletal pain: a comprehensive model. Man Ther. 2009 Oct;14(5):531-8. doi: 10.1016/j.math.2008.09.001. Epub 2008 Nov 21. PMID 19027342
- [Background] Lozano Lopez C, Mesa Jimenez J, de la Hoz Aizpurua JL, Pareja Grande J, Fernandez de Las Penas C. Efficacy of manual therapy in the treatment of tension-type headache. A systematic review from 2000-2013. Neurologia. 2016 Jul-Aug;31(6):357-69. doi: 10.1016/j.nrl.2014.01.002. Epub 2014 May 22. English, Spanish. PMID 24856370
- [Background] Schmid A, Brunner F, Wright A, Bachmann LM. Paradigm shift in manual therapy? Evidence for a central nervous system component in the response to passive cervical joint mobilisation. Man Ther. 2008 Oct;13(5):387-96. doi: 10.1016/j.math.2007.12.007. Epub 2008 Mar 3. PMID 18316238
- [Background] Shi X, Rehrer S, Prajapati P, Stoll ST, Gamber RG, Downey HF. Effect of cranial osteopathic manipulative medicine on cerebral tissue oxygenation. J Am Osteopath Assoc. 2011 Dec;111(12):660-6. PMID 22182951
- [Background] Morin CM, Belleville G, Belanger L, Ivers H. The Insomnia Severity Index: psychometric indicators to detect insomnia cases and evaluate treatment response. Sleep. 2011 May 1;34(5):601-8. doi: 10.1093/sleep/34.5.601. PMID 21532953
- [Background] Veqar Z, Hussain ME. Validity and reliability of insomnia severity index and its correlation with pittsburgh sleep quality index in poor sleepers among Indian university students. Int J Adolesc Med Health. 2017 Jan 7;32(1):/j/ijamh.2020.32.issue-1/ijamh-2016-0090/ijamh-2016-0090.xml. doi: 10.1515/ijamh-2016-0090. PMID 28063259
- [Result] Curtis BJ, Williams PG, Jones CR, Anderson JS. Sleep duration and resting fMRI functional connectivity: examination of short sleepers with and without perceived daytime dysfunction. Brain Behav. 2016 Sep 15;6(12):e00576. doi: 10.1002/brb3.576. eCollection 2016 Dec. PMID 28031999
- [Result] Jakel A, von Hauenschild P. Therapeutic effects of cranial osteopathic manipulative medicine: a systematic review. J Am Osteopath Assoc. 2011 Dec;111(12):685-93. PMID 22182954
- [Result] Hurley DA, Eadie J, O'Donoghue G, Kelly C, Lonsdale C, Guerin S, Tully MA, van Mechelen W, McDonough SM, Boreham CA, Heneghan C, Daly L. Physiotherapy for sleep disturbance in chronic low back pain: a feasibility randomised controlled trial. BMC Musculoskelet Disord. 2010 Apr 16;11:70. doi: 10.1186/1471-2474-11-70. PMID 20398349
- [Result] Levendowski DJ, Popovic D, Berka C, Westbrook PR. Retrospective cross-validation of automated sleep staging using electroocular recording in patients with and without sleep disordered breathing. Int Arch Med. 2012 Jun 25;5(1):21. doi: 10.1186/1755-7682-5-21. PMID 22726270
- [Result] Short NA, Allan NP, Raines AM, Schmidt NB. The effects of an anxiety sensitivity intervention on insomnia symptoms. Sleep Med. 2015 Jan;16(1):152-9. doi: 10.1016/j.sleep.2014.11.004. Epub 2014 Nov 25. PMID 25547037
- [Result] Jackowska M, Dockray S, Endrighi R, Hendrickx H, Steptoe A. Sleep problems and heart rate variability over the working day. J Sleep Res. 2012 Aug;21(4):434-40. doi: 10.1111/j.1365-2869.2012.00996.x. Epub 2012 Feb 7. PMID 22309485
- [Result] Toro-Velasco C, Arroyo-Morales M, Fernandez-de-Las-Penas C, Cleland JA, Barrero-Hernandez FJ. Short-term effects of manual therapy on heart rate variability, mood state, and pressure pain sensitivity in patients with chronic tension-type headache: a pilot study. J Manipulative Physiol Ther. 2009 Sep;32(7):527-35. doi: 10.1016/j.jmpt.2009.08.011. PMID 19748404
- [Result] Cutler MJ, Holland BS, Stupski BA, Gamber RG, Smith ML. Cranial manipulation can alter sleep latency and sympathetic nerve activity in humans: a pilot study. J Altern Complement Med. 2005 Feb;11(1):103-8. doi: 10.1089/acm.2005.11.103. PMID 15750368
- [Result] Miana L, Bastos VH, Machado S, Arias-Carrion O, Nardi AE, Almeida L, Ribeiro P, Machado D, King H, Silva JG. Changes in alpha band activity associated with application of the compression of fourth ventricular (CV-4) osteopathic procedure: a qEEG pilot study. J Bodyw Mov Ther. 2013 Jul;17(3):291-6. doi: 10.1016/j.jbmt.2012.10.002. Epub 2012 Nov 16. PMID 23768271